CLINICAL TRIAL: NCT05661266
Title: Investigating Eye-Movement Biomarkers of Disease Severity and Cognition in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Innodem Neurosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ETNA-subMS
Record Dates: First submitted 2022-12-02; First posted 2022-12-22 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort of MS patients with EDSS 0-8.0: Confirmed diagnosis of MS with an EDSS score ranging from 0 and 8.0.
  Interventions: Device: Eye-Tracking

INTERVENTIONS:
Device: Eye-Tracking — Eye-tracking technology and algorithms used to successfully capture and track eye movements using an electronic tablet and the embedded camera of the device.

SUMMARY:
The overarching goal of this research protocol is to acquire eye-tracking, cognitive, and disease-severity metrics in multiple sclerosis (MS) patients to further build up a database of MS patients and train a machine learning classifying algorithms to identify which eye-tracking metrics-or combination thereof-can serve as reliable markers of MS disease severity and cognitive status.

DETAILED DESCRIPTION:
This study will use a single group design in a cohort of MS patients. Eligible patients with MS will be selected and categorized based on their Expanded Disability Status Scale (EDSS) score. Patients eye movements will be captured using the patented eye-tracking technology at one single time point. In addition to the eye-tracking tests, patient phenotypes will be further detailed via brief functional and cognitive assessments using the EDSS, Brief International Cognitive Assessment for MS (BICAMS) and Multiple Sclerosis Functional Composite (MSFC). All patients will be required to participate in a single session.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Aged 18 years or older at the time of enrollment.
* Able to read in either French or English.
* Visual acuity of 20/100 in at least one eye (corrective glasses, contact lenses, surgery etc. are permitted)
* Confirmed diagnosis of MS with no signs of progressive increase in physical disability within the past six months.
* Neurological condition is medically stable during the study visit.

Exclusion Criteria:

* Evidence or medical history of psychiatric issues, which are known to also affect movements and oculomotor control.
* Presence of comorbid neurological conditions to avoid eye movement anomaly confounds (Strabismus, cranial nerve palsy, stroke-causing hemianopsia).
* Diagnosis of macular edema or other pre-existing ocular conditions that would prevent a participant from performing the eye movement assessments.
* Recent (less than three months from enrollment) start of, change of dose, or irregular use of, new prescription drugs known to influence ocular motor visual function, such as benzodiazepines, antipsychotics and anticonvulsants. Occasional use of benzodiazepines for medical procedures is permitted, at the investigator's discretion, but should not occur within a short time period prior to or during an eye movement assessment
* Diagnosis of Clinically Isolated Syndrome (CIS), Radiologically Isolated Syndrome (RIS) or Primary Progressive MS (PPMS).
* Patients who are currently experiencing a relapse or who have experienced a relapse within the last three months. A relapse is defined as appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must have been present for at least 24 hours and occurred in the absence of fever (< 37.5°C) or known infection.
* Patients who have been undergoing disease-modifying therapy for less than three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our target sample size for the MS group is 120. Eligible patients with MS will be selected and categorized based on their EDSS score.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Predictive power of eye-movement biomarkers (EMBs) for MS severity in relationship to Expanded Disability Status Scale (EDSS) | Day 1
  Estimate the extent to which EMBs can accurately predict MS severity (as assessed with the EDSS tool). The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.

SECONDARY OUTCOMES:
Predictive power of eye-movement biomarkers (EMBs) for cognitive status in relationship to the Symbol Digit Modalities Test (SDMT) as part of the Brief International Cognitive Assessment for MS (BICAMS). | Day 1
  The Brief International Cognitive Assessment for MS (BICAMS) is a battery of tests recommended by multiple sclerosis (MS) experts to monitor MS-related cognitive impairment, which includes the Symbol Digit Modalities Test (SDMT). The test presents a series of nine symbols, each paired with a single digit in a key at the top of a standard sheet of paper. Patients are asked to voice or write the digit associated with each symbol as rapidly as possible for 90 seconds. The test is scored on the number correct answers over the 90 second time span. A higher score represents lower levels of disability.
Predictive power of eye-movement biomarkers (EMBs) for cognitive status in relationship to the the California Verbal Learning Test-2 (CVLT2) as part of the Brief International Cognitive Assessment for MS (BICAMS). | Day 1
  The Brief International Cognitive Assessment for MS (BICAMS) is a battery of tests recommended by multiple sclerosis (MS) experts to monitor MS-related cognitive impairment, which includes the California Verbal Learning Test-2 (CVLT2). The test begins with the examiner reading a list of 16 words. Patients listen to the list and report as many of the items as possible. There is no instruction as to the order in which items are recalled. After recall is recorded, the entire list is read again followed by a second attempt at recall. Altogether, there are five learning trials. The reader will note that the 16-item list has words that conform to four semantic categories, in this case sports, vegetables, clothes, and tools. The test is scored on the total number of recalled items over the five learning trials. A higher score represents lower levels of disability.
Predictive power of eye-movement biomarkers (EMBs) for cognitive status in relationship to the Brief Visuospatial Memory Test-Revised (BVMT-R) as part of the Brief International Cognitive Assessment for MS (BICAMS). | Day 1
  The Brief International Cognitive Assessment for MS (BICAMS) is a battery of tests recommended by multiple sclerosis (MS) experts to monitor MS-related cognitive impairment, which includes the Brief Visuospatial Memory Test-Revised (BVMT-R). In this test, six abstract designs are presented for 10 sec. The display is removed from view and patients render the stimuli via pencil on paper manual responses. Each design receives from 0 to 2 points representing accuracy and location. Thus, scores range from 0 to 12. There are three learning trials, and the test is scored on the total number of points earned over the three learning trials. A higher score represents lower levels of disability.
Predictive power of eye-movement biomarkers (EMBs) for physical disability in relationship to the Timed 25-foot walk as part of the Multiple sclerosis functional composite (MSFC). | Day 1
  The Timed 25-Foot Walk is a quantitative measure of lower extremity function. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. The test is scored on the time taken to walk the two trials of the 25 feet walk. A higher score represents higher levels of disability.
Predictive power of eye-movement biomarkers (EMBs) for physical disability in relationship to the 9-Hole Peg Test (9-HPT) as part of the Multiple sclerosis functional composite (MSFC). | Day 1
  The 9-Hole Peg Test (9-HPT) is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and non-dominant hands are tested twice (two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand). The test is scored on the time taken to complete each trial for each hand. A higher score represents higher levels of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Genge Partners, Inc., Montreal, Quebec, Canada